CLINICAL TRIAL: NCT00351338
Title: Preoperative Nutritional Deficiencies in the Bariatric Surgery Patients
Brief Title: Nutritional Deficiencies in the Bariatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: chayas-HMO-CTIL
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2006-07

CONDITIONS: Morbid Obesity; Nutritional Deficiency
MeSH Terms: conditions — Obesity, Morbid; Malnutrition

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Although morbidly obese subjects have larger than regular caloric intake, there is evidence that they suffer from nutritional deficiencies at a higher rate than the general population, probably because they eat mostly "unhealthy food."

ELIGIBILITY:
Inclusion Criteria:

* All morbidly obese subjects who are surgery candidates

Exclusion Criteria:

* Previous bariatric operations

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Keidar, MD, Principal Investigator — Hadassah Medical Organization Israel
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel